CLINICAL TRIAL: NCT02802267
Title: Efficacy Study of Inecalcitol in Combination With Decitabine in Acute Myeloid Leukemia Patients Unfit for Standard Chemotherapy
Brief Title: Efficacy Study of Inecalcitol With Decitabine in Acute Myeloid Leukemia Patients Unfit for Standard Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hybrigenics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICT8
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — inecalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- inecalcitol (Experimental): Two tablets of Inecalcitol 2mg each (total 4mg) taken orally every other day.
  Interventions: Drug: Inecalcitol
- placebo (Placebo Comparator): Two tablets of placebo 2mg each (total 4mg) taken orally every other day
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Inecalcitol — vitamin D receptor agonist
  Arms: inecalcitol
Drug: Placebo Oral Tablet — placebo
  Arms: placebo

SUMMARY:
Evaluate the effect of the addition of inecalcitol to decitabine treatment on overall survival in previously untreated AML patients aged 65 years or more who are randomly assigned to receive decitabine with or without inecalcitol.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged 65 to < 75 years with at least one non severe comorbidity ie disease or syndrome with mild to moderate clinical or diagnostic observations or lab abnormalities which could increase the risk of toxicity and/or early death of intensive chemotherapy in the opinion of the investigator and are not contra-indicated for non-intensive chemotherapy.

or ≥ 75 years with or without any comorbidity at the time of the informed consent signature;

• Newly diagnosed, untreated de novo or secondary AML according to WHO classification;

Exclusion Criteria:

* Prior or current treatment with chemotherapy for any myeloid disorder (excluding hydroxyurea) or radiotherapy for extramedullary involvement within 2 weeks of randomization;
* Prior treatment with decitabine, azacitidine, or cytarabine;
* Prior malignancies for 5 years with exception of basal cell, squamous cell carcinoma of the skin, or carcinoma " in situ " of the cervix or breast;
* Chronic myelogenous or acute promyelocytic leukaemia;
* Known CNS involvement;
* Patient eligible to bone marrow or stem cell transplant;
* WBC ≥ 30.000/mm3;
* Impaired renal function with Creatinine clearance < 30 mL/min/1.73m² according to the MDRD formula;
* Serum bilirubin ≥ 2.5 x ULN and/or AST and/or ALT ≥ 2.5 x ULN (upper limit of normal value);
* Calcemia ≥ 2.65 mmol/L (106 mg/L) at screening assessment (corrected with albuminemia);
* History of diseases known to be associated with calcium disorders: ongoing hyperparathyroidism, sarcoidosis….;
* Presence or history of symptomatic kidney stones in the last 5 years;
* Hypersensitivity to any of the excipients of decitabine (Potassium dihydrogen phosphate (E340) ; Sodium hydroxide (E524) ; Hydrochloric acid (for pH adjustment) or to the excipient of inecalcitol tablets (lactose);
* Current use of drugs known to influence serum calcium (such as thiazide diuretics, teriparatide, calcitonin and multivitamin supplements containing > 400 IU of vitamin D or calcium);
* Current use of digitalis;
* Current use of drugs which could influence bioavailability of inecalcitol (such as magnesium-containing antacids, bile-resin binders);
* Use of any other experimental drug or therapy or vitamin D supplementation within 4 weeks of randomization;
* Known HIV;
* Patients who are eligible for intensive induction therapy with curative intent;
* Refractory congestive heart failure;
* Active infection resistant to anti-infective therapy;
* Documented pulmonary disease with DLCO ≤ 65% or FEV1≤ 65%, or dyspnea at rest or requiring oxygen, or any pleural neoplasm or uncontrolled lung neoplasm;
* Liver cirrhosis Child B or C or acute viral hepatitis;
* Current mental illness requiring psychiatric hospitalization, institutionalization or intensive outpatient management, or current cognitive status that produces dependence (as confirmed by the specialist) not controlled by the caregiver;
* Uncontrolled neoplasia;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Dufour-Lamartinie, MD, Principal Investigator — Hybrigenics Corporation
Locations (8):
- United States (7):
  - Scripps Health, San Diego, California
  - Georgia Cancer Center-Augusta University, Augusta, Georgia
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Duke Cancer Institute, Duke Univ Medical Center, Durham, North Carolina
  - University of Texas; M D Anderson Cancer Center, Houston, Texas
  - ProHealth Care Inc, Waukesha, Wisconsin
- Necker Hospital- APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No